CLINICAL TRIAL: NCT05833425
Title: Is Respiratory Muscle Strength, Peripheral Muscle Strength and Postural Control Affected in Adolescent Idiopathic Scoliosis?
Brief Title: Is Respiratory Muscle Strength, Peripheral Muscle Strength and Postural Control Affected in Scoliosis?
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BVUsyildirim02
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Adolescent Idiopathic Scoliosis; Respiratory Muscle Strength; Peripheral Muscle Strength; Postural Control
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scoliosis group: In this study, an evaluation form including demographic and clinical characteristics, respiratory muscle strength measurement, quadriceps muscle strength measurement with electronic hand dynamometer, hand grip strength with dynamometer and postural stability assessment with Biodex Balance System® will be applied to all scoliosis adolescent.
  Interventions: Device: Respiratory Pressure Meter (MicroRPM)
- Healthy group: In this study, an evaluation form including demographic and clinical characteristics, respiratory muscle strength measurement, quadriceps muscle strength measurement with electronic hand dynamometer, hand grip strength with dynamometer and postural stability assessment with Biodex Balance System® will be applied to all healthy adolescent.
  Interventions: Device: Respiratory Pressure Meter (MicroRPM)

INTERVENTIONS:
Device: Respiratory Pressure Meter (MicroRPM) — Peripheral muscle strength, respiratory muscle strength and postural controls of all adolescents will be evaluated. The values of the scoliotic and healthy groups will be compared.
  Other Names: Biodex Balance System®

SUMMARY:
The vertebral column is a structure that transfers the weight of the head and torso to the lower extremity, provides trunk movements and protects the spinal cord.A three dimensional deformity involving lateral flexion of the vertebrae in the frontal plane at 10 ° and above, including axial rotation and physiologic flexion (hypokyphosis) components in the sagittal plane, is defined as scoliosis. Adolescent idiopathic scoliosis (AIS) is a type of idiopathic scoliosis that occurs in the period from the onset of puberty (up to 10 years) until the closure of growth plates.

Scoliosis is caused by postural, balance and neuromotor disorders as a primary cause of impaired sensory integrity, proprioceptive feedback deficits, secondary lung problems, organ disorders and pain. Children with adolescent idiopathic scoliosis have inadequate respiratory function. At the same time, these children show muscle weakness in certain parts of the body.

The aim of this study is to compare young adolescents with scoliosis with their healthy peers and examine whether respiratory muscle strength, peripheral muscle strength and postural control are affected.

ELIGIBILITY:
Inclusion Criteria:

* Individuals agreeing to participate in the study
* In the age range of 10-20
* Patients with scoliosis with a Cobb angle of 15-40 degrees measured on X-Ray

Exclusion Criteria:

* Surgical operation in the last 3 months
* Having mental, communicative and behavioral disorders that may cause problems understanding commands and questions or performing exercises.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: It was calculated that at least 36 patients in total, 18 patients in the scoliosis and healthy groups, should be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | Baseline
  Respiratory muscle strength will be made with a portable, electronic intraoral pressure measuring device.
Peripheral Muscle Strength | Baseline
  Peripheral muscle strength will be performed using an electronic dynamometer.
Postural Control | Baseline
  Postural Stability and Balance will be evaluated with the Biodex Balance System®.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüp, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided